CLINICAL TRIAL: NCT03488095
Title: Behavior Changing Intervention for Smokeless Tobacco and Betel Quid Use in Adolescents: A Cluster-Randomized Trial
Brief Title: Behavior Changing Intervention for Smokeless Tobacco and Betel Quid Use in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Prof. Dr. Azmina Hussain, Professor, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DUHS/DR-O/2016/116
Record Dates: First submitted 2018-03-21; First posted 2018-04-04 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Oral Cavity Carcinoma
Keywords: Tobacco, smokeless, chewing, betel quid
MeSH Terms: conditions — Mouth Neoplasms | interventions — 2-benzylidene-3-(cyclohexylamino)-2,3-dihydro-1H-inden-1-one

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavior changing intervention (Other): Thirty minutes behavior counselling (PPT.) to experimental group. BCI for SLT and BQ Use in Adolescents: A CRT
  Interventions: Behavioral: BCI for SLT and BQ Use in Adolescents: A CRT
- Control Cluster (No Intervention): No thirty minutes behavior counselling (PPT.) to control group

INTERVENTIONS:
Behavioral: BCI for SLT and BQ Use in Adolescents: A CRT — BCI for SLT and BQ Use in Adolescents: A CRT is aimed towards changing Adolescenst behaviors regarding their SLT and BQ use to as to reduce Oral cancer Burden within population because of this.
  Arms: Behavior changing intervention

SUMMARY:
Smokeless tobacco (SLT) is a known risk factor for Oral, Pharyngeal and Esophageal carcinoma. Three-quarters global SLT consumption is among the South Asian Population. The habit of SLT chewing commences at a very young age which has an underpinning of socio-cultural dimension in South Asian population which perhaps due to its more addictive potential, has more dependency. Youth also perceives SLT as a part of confectionery, which is socially served in South Asian ceremonies. There exists very little or no evidence regarding efficacy of SLT cessation interventions in this population. Most of the existing interventions are based in western world with little or no cultural sensitivities pertinent to South Asia. In this study, a culturally rooted behavior changing intervention (BCI) to alter SLT use prevalence, perceptions pertinent to the deleterious effects of SLT use in the etiology of oral cancers and help youth quit SLT in Karachi, Pakistan.

Baseline demography and SLT use prevalence will be ascertained among 11-16-year-old school going children from both government and private schools. Multi stage cluster sampling will randomly recruit forty clusters (schools) from within 6 districts of Karachi, which will then be divided into intervention and control groups (clusters) using block randomization based on proportionate number of each school type present (Government and Private).

Both groups' participants will complete all questionnaires pre and post intervention as described elsewhere and will also undergo screening for oral cancer and oral potentially malignant lesions (OPMLs). Students in intervention cluster will be given BCI and printed pamphlets along with a gift pack (reminder for SLT quit, a branded tooth paste and a tooth brush) while students in control cluster will only differ in that they will not be exposed to BCI.

BCI was designed after reviewing literature and consulting specialist group for all untoward effects of SLT use in Oral Cavity that have a potential of transforming into oral carcinoma.

A follow up after 12 weeks will be conducted to re-assess their SLT use prevalence, perceptions regarding hazardous effects of SLT use in oral cavity, dependency on SLT and success in quit (among users in both groups), and perception regarding warning labels on SLT product packet

DETAILED DESCRIPTION:
In lieu of the increasing disease burden of oral cancer in South Asian countries due to increasing popularly fashionable SLT consumption; the objective is to develop (i) a BCI pertinent to socio-cultural aspect for South Asian SLT users, followed by (ii) assessing its efficacy in changing perception and dependency regarding SLT use in high risk group of 11-16 years old school going children of Karachi of both private and public sector schools.

It is also aimed to deconstruct the BCI to establish which components of our BCT are more useful in making an intervention most efficient by using sub-indices of fidelity index to assess the adherence and quality of each component of intervention. Each component will be scored using fidelity index by a neutral trained listener each time intervention is delivered by a trained personnel.

Quantitatively, the objectives of the study are to:

i. measure SLT/ or BQ use prevalence amongst adolescents of 11-16 years ii. assess the reasons behind their use of SLT/ or BQ in users (both intervention and control clusters) by using Reasons for Betel Quid Chewing Scale (RBCS).

iii. evaluate the dependency on SLT/ or BQ in users (both intervention and control clusters) using Fagerstörm Tobacco and Nicotine Dependency scale for Smokeless Tobacco (FTND-ST) and Betel Quid Dependency by using Betel Quid Dependency Scale (BQDS).

iv. assess perceptions of adolescents (both intervention and control clusters) regarding ill effects of SLT/ or BQ use in oral cavity causing oral cancer and OPMLs.

v. assess the perception of adolescents regarding oral cancer picture of SLT/ or BQ product pack in cessation of its use with the help of Behavior Changing Intervention in intervention cluster and a questionnaire item in control cluster.

vi. evaluate each component of Behavior Changing Intervention in its efficacy by using fidelity index and self-perceived efficacy by participants of intervention cluster.

This study will be conducted at government and private schools of Karachi as schools have the maximum probability of engaging focused age group of mixed ethnicity, religion, different cultures and different socio-economic strata of the population. Also, these young individuals spend a substantial number of their waking hours in school thus they are easily approachable globally without needing to delineate or be reliant on families(41).

With a population of approximately 24 million, Karachi is the largest city of Pakistan(42). Karachi City government has divided the city into six (6) districts in 2013 with each district being further divided into administrative towns of total 18 in number(43).

Multi stage cluster sampling will be done. Out of six districts, 26 clusters (secondary schools) will be randomly selected proportionate to the number of each school type (ensuring equal participation of government and private schools). The students of 11-16 years of age, studying in grade VI - Grade X will be randomly recruited. Complete lists of all private and government schools of Karachi have been arranged by requesting respective Directors (Appendix 6). If any randomly selected school declines to participate than another school will be randomly selected from the same district; also, a government school will be selected if government school will decline and vice versa. Fifty-100 students per school will be randomly included in the study. Depending upon the size of each class, students will be randomly selected from each of the secondary classes present on the day of our visit till a total number of 50-100 is reached.

This will therefore summit a total sample size of 2200 that may be considered representative of the 11-16 year adolescents of Karachi as Global Youth Tobacco Survey conducted in Karachi, Pakistan in 2008 enrolled 720 individuals of 13-15 years for comprehensive tobacco control program(44).

Students of younger or older age group than mentioned already will be excluded and students who already are undergoing treatments for Oral Cancer will be excluded.

For recruitment purposes, investigators will contact principals of selected schools (both government and private) to provide them with details regarding the intervention, its merits and efficacy, and will request for their inclination to participate in the trial. If any selected school refuses to participate then another school of same profile will be sent an invitation.

Schools' heads will then be requested to send consent forms (will be provide to schools) to the parents along with a covering letter in which they will be provided with all relevant details regarding intervention and will be encouraged to contact principal investigator via a text on given contact number who will then call parents to respond to all queries since principal investigator does not have toll-free number(33).

Parents will be requested to sign an acceptance or refusal on the form and sent it back to school by a specific decided date.

After 12 weeks, a follow up visit will ensue to:

1. Re-assess their perceptions regarding SLT/or BQ use in users and non-users of both intervention and control clusters.
2. Re-assess their dependency on SLT/or BQ in users of both intervention and control clusters.
3. Re-evaluate their perceptions (of users and non-users of intervention cluster) regarding warning labels on SLT/or BQ product packet
4. Collect their quit calendars to assess quit from users of both intervention and control clusters, and
5. Collect perceived efficacy of each component of BCI that helped them quit, attempt to quit or change perceptions from all users and non-users of intervention cluster to assess efficacy of each component of BCI.

Any differences in outcome based on BCI will be assessed and documented between two arms of cluster-randomized trial.

The change in perceptions if at all, after four weeks, regarding imprinting of pictorial warning labels on SLT packaging will help us in recommending its implementation at National level to curb SLT use.

ELIGIBILITY:
Inclusion Criteria:

• 11-16 years school going children with NO diagnosed oral cancer

Exclusion Criteria:

* Students younger or older than mentioned ages
* Diagnosed Oral Cancer patients

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2200 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Changing perceptions regarding SLT and BQ use | 3 months
  modified Global Youth Tobacco Survey will be used to assess the perceptions of adolescents

SECONDARY OUTCOMES:
prevalence of SLT and BQ use in 11-16-year-old | 3 months
  modified Global Youth Tobacco Survey will be used
Quit/quit attempts by the participants | three months
  modified Global Youth Tobacco Survey will be used
prevalence of OPMLs in the users of SLT and BQ | three months
  modified Global Youth Tobacco Survey will be used
perceptions regarding warning labels on SLT and BQ product pack | three months
  modified Global Youth Tobacco Survey will be used

CONTACTS AND LOCATIONS:
Overall Officials: Kashif Sahfique, PhD, Study Chair — Dow University of Health Sciences
Locations (1):
- DOW University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
once avaialble, it will be shared
Supporting Information: SAP
Time Frame: when study results are published
Access Criteria: confidentiality will need to be maintained

REFERENCES:
- [Derived] Hussain A, Zaheer S, Shafique K. School-based behavioral intervention to reduce the habit of smokeless tobacco and betel quid use in high-risk youth in Karachi: A randomized controlled trial. PLoS One. 2018 Nov 2;13(11):e0206919. doi: 10.1371/journal.pone.0206919. eCollection 2018. PMID 30388182